CLINICAL TRIAL: NCT01669109
Title: Hatha Yoga for Patients With Colorectal Cancer - a Randomized Controlled Trial
Brief Title: Hatha Yoga for Patients With Colorectal Cancer
Acronym: YoCo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Postdoctoral fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-4957-BO
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Neoplasms
Keywords: Yoga; Colorectal Neoplasms; Quality of Life; Randomized Controlled Trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hatha yoga (Experimental): * 10 weeks of Hatha yoga, designed for patients with colorectal cancer, as a group intervention
  * 1 weekly class (90 minutes)
  Interventions: Behavioral: Hatha yoga
- Usual care (No Intervention): Patients continue their self-directed usual care

INTERVENTIONS:
Behavioral: Hatha yoga
  Arms: Hatha yoga

SUMMARY:
Hatha Yoga is a traditional practice that encompasses aerobic exercise, breathing techniques, and meditation. It is used in India since centuries to improve well-being and cope with diseases and is gaining more and more interest in Europe and the US. While studies have demonstrated benefits of Hatha Yoga for patients with breast cancer, no studies on patients with colorectal cancer are available yet. The purpose of this study is to investigate the effect of Hatha Yoga in patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer
* UICC stage I-III
* between 2 and 48 months post-surgery
* age at least 18 years
* physical and cognitive ability to follow the yoga intervention

Exclusion Criteria:

* UICC stage IV
* further active oncological diseases
* diagnosed and pharmacologically treated psychiatric disorder except for cancer-related depression or adjustment disorder
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Week 10
  Functional Assessment of Cancer Therapy - Colorectal Cancer (FACT-C)

SECONDARY OUTCOMES:
Health-related quality of life | Week 22
  - Functional Assessment of Cancer Therapy - Colorectal Cancer (FACT-C)
Fatigue | Week 10, week 22
  Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
Anxiety, depression | Week 10, week 22
  Hospital Anxiety and Depression Scale (HADS)
Sleep quality | Week 10, week 22
  Pittsburgh Sleep Quality Index (PSQI)
Safety | Week 0-22
  Number and severity of adverse events
Spiritual well-being | Week 10, week 22
  - Functional Assessment of Chronic Illness Therapy - Spirituality (FACIT-Sp)

OTHER OUTCOMES:
Body awareness/bodily dissociation | Week 10, week 22
  * Scale of Body Connection (SBC)
  * Used in mediation analysis
Body efficacy expectation | Week 10, week 22
  * Body Efficacy-Expectation Scale
  * Used in mediation analysis
Qualitative Interviews | Week 11

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Department of Internal and Complementary Medicine, Immanuel Hospital Berlin, Berlin
  - Department for Internal and Integrative Medicine, Essen-Mitte Clinics, Essen

REFERENCES:
- [Derived] Cramer H, Pokhrel B, Fester C, Meier B, Gass F, Lauche R, Eggleston B, Walz M, Michalsen A, Kunz R, Dobos G, Langhorst J. A randomized controlled bicenter trial of yoga for patients with colorectal cancer. Psychooncology. 2016 Apr;25(4):412-20. doi: 10.1002/pon.3927. Epub 2015 Jul 29. PMID 26228466